CLINICAL TRIAL: NCT06424015
Title: Effect of Insulin and Insulin Pulses on Fasting Glucagon Secretion and on Glucose Metabolism in Subjects Without Type 2 Diabetes
Brief Title: Insulin and Insulin Pulses During Fasting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24-002631
Record Dates: First submitted 2024-05-13; First posted 2024-05-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: PreDiabetes
Keywords: insulin secretion; glucagon secretion; endogenous glucose production; glucose disappearance
MeSH Terms: conditions — Prediabetic State | interventions — soybean oil, phospholipid emulsion; Heparin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralipid and heparin (Active Comparator): Between 0600 (-180 min) and 1300 (240 min) Intralipid (20%, 0.011ml/kg/min; Baxter, Healthcare, Deerfield, IL) and heparin (200 units prime, 0.2 unit/kg/min continuous) will be infused to induce acute insulin resistance.
  Interventions: Other: Intralipid and heparin
- Saline (Placebo Comparator): Between 0600 (-180 min) and 1300 (240 min) saline will be infused
  Interventions: Other: Saline

INTERVENTIONS:
Other: Intralipid and heparin — Intralipid (20%, 0.011ml/kg/min; Baxter, Healthcare, Deerfield, IL) and heparin (200 units prime, 0.2 unit/kg/min continuous) will be infused to induce acute insulin resistance
  Arms: Intralipid and heparin
Other: Saline — Saline will be infused
  Arms: Saline

SUMMARY:
Fasting hyperglycemia contributes disproportionately to nonenzymatic glycosylation and the microvascular complications of type 2 diabetes. However, little is known about the regulation of glucose concentrations in the fasting state relative to what is known about the postprandial state. The proposed experiment is part of a series of experiments designed to establish how glucagon and insulin interact with their receptors to control fasting glucose in health and in prediabetes.

DETAILED DESCRIPTION:
Decreased insulin action increases glucagon concentrations. In rodents, insulin signaling restrains glucagon secretion. It is unclear if this is the case in all (subtypes of) prediabetes. Impaired hepatic insulin action exacerbates glucagon's effects on endogenous glucose production. Also, insulin resistance in the β-cell impairs negative feedback inhibition of insulin secretion. This leads to hyperinsulinemia in rodents and humans. How these variables interact is unknown. This experiment will determine how insulin variably regulates fasting glucagon (and insulin) secretion directly, or indirectly, in prediabetes.

The inability of the proinsulin to insulin ratio to reliably predict β-cell integrity, endoplasmic reticulum stress and β-cell function has led to the identification of novel markers of β-cell health. In addition, the relationship of glucagon and insulin pulses will be quantified. Preliminary data shows that there is heterogeneity in these relationships even in normal fasting glucose. Th experiment will also determine how islet hormone / glucose crosstalk and pulse characteristics contribute to prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* people with normal or impaired fasting glucose and normal or impaired glucose tolerance

Exclusion Criteria:

1. HbA1c > 6.5%
2. BMI ≥ 35 Kg/M2
3. Use of any glucose-lowering agents including metformin or sulfonylureas.
4. For female subjects: positive pregnancy test at the time of enrollment or study
5. History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
6. Active systemic illness or malignancy.
7. Symptomatic macrovascular or microvascular disease.
8. Hematocrit < 35%

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Suppression of Endogenous glucose production (EGP) by insulin | The rate of EGP at 240 minutes (end of study) expressed as a percentage of fasting EGP (at the start of the study i.e.: 0 minutes.
  comparison of EGP in people with IFG vs NFG in response to insulin infusion
Insulin pulse orderliness | Approximate Entropy (ApEn) will be calculated from the insulin concentrations observed every 2 minutes between -45 and 0 minutes
  comparison of Insulin pulse orderliness measured by approximate entropy in people with IFG vs NFG

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that will be preserved and shared include results of screening labs, immunoassay data and glucose turnover data. In addition, we will share the study protocol, statistical analysis plan, a data dictionary and anonymization guidance (methodology to anonymize data).In addition to the patient-level data, the metadata, data dictionary, statistical analysis plan, and final protocol will be shared. The sharing of the data dictionary, statistical analysis plan and final protocol with amendments will enable researchers to understand how the data was collected and to correctly interpret the data for future secondary analysis. The final patient level dataset will include demographics as well as screening data and primary and secondary outcomes.We plan to share datasets resulting from the proposed studies in Vivli, a non-profit institution that supports the Vivli repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data shared will be archived and available on the platform for request by researchers for a minimum of 10 years after contribution. Data will be made accessible no later than the time of our associated publication or the end of the grant period (whichever comes first). On an ongoing basis, Vivli evaluates its data holdings regarding maintaining access and reserves the right to discontinue the distribution of a data collections when deemed appropriate. When materials are deaccessioned, the data are no longer publicly accessible at Vivli, they may still be preserved in Vivli's storage vault. Because digital files are assigned a persistent digital object identifier (DOI), the study description is still available to view, but is not searchable through Vivli.
Access Criteria: The data being shared is human data from clinical trials and therefore a higher level of protection is required. Access to this data will be controlled by a managed access process whereby access is provided only after approval. Data will be controlled access with the General Research Use Data Use Limitation, as allowed by the informed consent and the institutional certification.